CLINICAL TRIAL: NCT03667079
Title: Integrating Community-directed Interventions to Eliminate Neglected Tropical Diseases Caused by Soil-transmitted Helminth Infections and Rabies in Tanzania
Brief Title: Integrating Community Interventions to Eliminate Neglected Tropical Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: University of Glasgow (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Felix Lankester, Research Associate Professor, Washington State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 14674-001
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Rabies in Animals; Worms; Intestine
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: Villages were allocated to one of three treatment arms: in Arm 1 villages people received deworming treatment and dogs rabies vaccination through an integrated delivery; in Arm 2 villages only deworming of people occurred; in Arm 3 only dog vaccination occurred. After the study, Arm 2 and 3 villages received rabies vaccination and deworming, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Integrated (Experimental): Intervention 'integrated delivery of deworming and vaccination' will be delivered to this arm of the study
  Interventions: Other: integrated delivery of deworming and vaccination
- Deworming only (Active Comparator): Intervention 'Mass deworming only' will be delivered to villages in this arm of the study
  Interventions: Other: Mass deworming only
- Rabies vaccination only (Active Comparator): Villages assigned to this arm received mass vaccination of dogs against rabies only
  Interventions: Other: Mass vaccination of dogs

INTERVENTIONS:
Other: integrated delivery of deworming and vaccination — integrated delivery of mass drug administrations, one targeting humans (deworming) and one targeting animals (rabies vaccination)
  Arms: Integrated
Other: Mass deworming only — Delivery of mass deworming to people only
  Arms: Deworming only
Other: Mass vaccination of dogs — Delivery of mass vaccination of dogs only
  Arms: Rabies vaccination only

SUMMARY:
The overarching goal of this project is the elimination of two neglected tropical diseases (NTD):

soil-transmitted helminthiasis and rabies. The specific objective of this pilot study was:

To determine whether the integrated delivery platform improved the cost-effectiveness and coverage of MDA targeting STH and rabies;

The investigators integrated two public health initiatives: 1) a mass drug administration (MDA) effort to eliminate neglected tropical diseases (NTD) caused by soil-transmitted helminths (STH), with 2) a community-valued mass dog rabies vaccination (MDRV) intervention to eliminate human and animal rabies, also a priority NTD of the World Health Organisation. The goal of MDA efforts targeting STH is to reduce worm burdens to very low levels below which self-sustaining transmission, and the public health consequences of STH, cease. Existing school-based delivery programs fail to reach all affected age groups, however, which results in ineffective coverage levels and persistence of STH. The goal of MDRV is to immunize 70% of dog populations, after which canine-mediated rabies is eliminated. MDRV programs are typically very popular, with all human age groups participating. The objectives of this project were to determine whether supplementing a strictly school-based MDA NTD control program with a community-wide strategy that is coupled to an MDRV program will result in a synergism that (a) improves coverage, reach and cost-effective delivery of MDA targeting STH and (b) improves coverage and cost-effective delivery of dog vaccination. To achieve this, research activities, comprised of post-intervention household questionnaire surveys, were carried out. In addition detailed cost data was collected.

DETAILED DESCRIPTION:
The study was carried out in the Ngorongoro District, Tanzania inhabited by semi-nomadic Maasai people. The remote area was chosen because MDRV and MDA are carried out annually in the region as separate programs. The MDA program delivers twice yearly deworming treatment to every primary school and is coordinated by the District Medical Office (DMO). The MDRV program vaccinates dogs annually and is coordinated by the District Veterinary Office. The MDA and MDRV carried out in this study constituted one cycle of the established MDA and MDRV in the target villages. The study took place between February and October 2016, however activities were suspended during the rainy season to avoid inclement weather from affecting participation.

The study focused on 24 villages. The target villages were located within the eight wards immediately surrounding the district's administrative centre and were selected through convenience. Each of the 24 villages were randomly assigned to one of three arms: i) Arm A (n = 8) received both MDA and MDRV; ii) Arm B (n = 8) received MDA only; iii) Arm C (n = 8) received MDRV only. All villages were equally likely to be assigned to each arm. As per the established MDA and MDRV programs, a nurse from the DMO and two village-based community health workers carried out the MDA whilst a rabies field team (a veterinarian, two field staff and a ward-based person) delivered the MRDV. STH and / or rabies awareness information was provided to respondents in the form of verbal disease avoidance advice.

Villages in this region cover a large area, and all are divided into sub-village units. Each intervention ('event') was delivered at the level of the sub-village using a 'central-point' strategy, which required villagers to travel from their homes to the central-point event to receive treatment. Village leaders estimated that hosting each sub-village event for one day would provide sufficient time for villagers to attend. Consequently each event was scheduled to last for one day, and the number of days the team(s) spent in each village equalled the number of sub-villages.

Arm A events comprised an MDA and a MDRV clinic hosted concurrently, while Arm B and Arm C events comprised only one clinic (MDA or MDRV, respectively). For Arm A villages, the MDA and MDRV delivery teams travelled together in one vehicle and set up the clinics close to each other. For Arm B and C villages, the MDA and MDRV teams travelled separately.

In order to allow comparison of the MDA with school-based delivery (second objective) the events were all hosted during the school term. In sub-villages with a primary school, the clinics were positioned outside the school grounds, whilst in sub-villages that did not have a primary school the clinics were located in a central location.

To inform each community of the event, a village-wide meeting was convened one week before. Key information provided at the meeting included STH and / or rabies awareness information and the importance of controlling these conditions through MDA and MDRV, the date of each clinic, that treatment would be given free of charge, and that people and dogs of all ages were invited to attend. On the Sunday prior to a village event, a motorbike rider with a loudspeaker drove around each village announcing the event details. Additionally the DMO informed the head teacher of each primary school of the date that the event would be convened outside of the school grounds. At 0830 hours the clinic(s) would be set up in the predetermined location and the treatment teams would wait for villagers to arrive. People coming to the MDA clinic were registered and research data collected. Following this, children between 12 and 59 months were given an oral dose of mebendazole (500mg) and vitamin A (100,000 IU), whilst people over 59 months were given an oral dose of albendazole (400mg). Following arrival and registration at the MDRV clinics, dogs were vaccinated (Nobivac Rabies®, MSD Animal Health, Boxmeer, Netherlands), a collar placed around the neck and water-soluble purple coloured paint was applied to both flanks. People attending the combined clinic (Arm A) who had also brought dogs were instructed to visit the MDRV clinic after receiving deworming treatment. The events ended at 1630 hours.

Household participation and coverage - community perceptions and knowledge:

A post-intervention household questionnaire survey (HQS) targeting 30 randomly selected households per village (stratified across sub-villages) was carried out within one week of each intervention to determine the proportion of households, people and dogs that attended the clinics. No households declined to participate, however if the family were not at home the team moved onto the next household.

Coverage of school-aged children and others:

To calculate the percentage of treated primary school age children (7 - 13 years) that were enrolled or not in school, or were attending or not attending school on the day of the clinic, every person treated was asked whether they were enrolled and attending primary school that day and, if they attended primary school, which primary school they attended. Every participant was also asked their age, which allowed analysis of other age groups treated.

Chi squared tests were used to determine whether household participation and coverage were impacted by delivery strategy. A logistic regression model (logit family) was used to determine whether the proportion of children enrolled in primary school in each village was dependent on the presence of a school.

Comparison with the national school-based deworming program:

To determine whether delivery strategy and clinic location (outside of school grounds with the whole community invited (this study) or within the schools with treatment given only to enrolled school children (NSDP)) impacted the number of school children that received deworming treatment, a paired comparison at ten village primary schools was made. To allow comparison, the number of primary school children treated in the previous NSDP round of deworming treatment was obtained for each of the ten schools from the Ngorongoro District NTD Coordinator and compared with the number of registered children treated in this study in the same schools.

A generalized linear mixed model, with 'school name' as a random effect, was used to compare the proportion of primary school children treated by the NSDP and this study in each comparison school.

Administration and delivery costs:

Clinic administration and delivery (A&D) costs were collected for all 24 villages, including variable costs (per dose delivered, by dose type) and fixed costs (per clinic, by clinic type). Expense categories included: Advertising, Equipment, Incentive payments to village leaders, Labour Costs (team salaries and wage labour for local help), Living (lodging) Allowance, Per Diem for the team, Meeting Costs, Vehicle Fuel, Repairs and Service, Communication (telephone credits), and Other. Other included a variety of miscellaneous costs that do not fit under any other category, such as incidental taxi and transportation costs and team health treatment. Costs attributable to research-related activities were not included in A&D costs. Indirect costs (time, foregone opportunities) borne by households to attend the event (described above) were not included in A&D costs. For accounting purposes, fixed costs not attributable to a specific clinic type were allocated equally across all events. Fixed costs attributable to either MDRV or MDA were attributed equally across all rabies or deworming events, respectively. Because there were two clinics for each Arm A event, the unattributable fixed cost per clinic was half that of Arm B and C. Variable costs per clinic were calculated as per-dose purchase costs multiplied by the number of doses delivered. Per-dose purchase costs were $0.021 (44 Tanzanian Shillings [Tsh]) per deworming dose and $0.26 (520 Tsh) per rabies vaccination. The exchange rate for cost calculations was 2,100 Tsh per U.S. Dollar, approximately the exchange rate that prevailed from mid-2015 through 2016.

The average cost per dose (A&D) was calculated in two ways. Method 1 calculates the total cost over all clinics (by clinic type and Arm) divided by the total number of doses delivered (by clinic type and Arm), and represents the aggregate cost per dose for a given clinic category. Method 2 calculates cost per dose on a per clinic basis, and then averages over all clinics. Both methods provide valid measures of cost per dose (A&D), but provide different estimates, because the average of a ratio (Method 2) is not equivalent to the ratio of averages or totals (Method 1). Method 1 is useful as an aggregate measure over all clinics, but cannot be used to test for statistical differences across clinic categories because it is not calculated on a per clinic basis. Method 2 allows testing for statistical differences across clinic types, but represents a summary statistic for clinic-level cost per dose measure rather than an aggregate measure.

Two-sample parametric and non-parametric tests were used to test for differences in cost per dose between Arms A and B, and Arms A and C.

Travel time to attend clinics:

To understand which mode of transport was most commonly used, respondents were asked how they travelled to the clinic (foot, carried (e.g. infants), bike, car, etc.). To estimate the mean time (t ̅_1) a respondent took attending a combined or single event, respondents were asked how long it took in minutes to reach the events. In addition, the mean amount of time a respondent spent at a clinic (t ̅_2) and, for the integrated delivery (Arm A) the mean time spent travelling between the two clinics (t ̅_3), was measured. These estimates were then used to compare the overall time spent attending single and integrated events. To estimate the overall time a respondent spent attending a single clinic (Arm B or C, or Arm A if no dog was brought for vaccination) (T_s) we multiplied the mean travel time by two (for the out and return journey) and added the mean time spent at a clinic:

T_s=(t ̅_1 × 2)+ t ̅_2.

To estimate the mean time a respondent spent attending a combined clinic (Arm A) (T_c ) we multiplied the mean travel time by two and added the mean time spent at a clinic (multiplied by two for deworming and dog vaccination) and the time spent travelling between the two clinics:

T_c=(t ̅_1× 2)+(t ̅_2× 2)+ t ̅_3.

ELIGIBILITY:
Inclusion Criteria:

* All healthy non pregnant people

Exclusion Criteria:

* Children attending clinics alone
* Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28143 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of people in each village receiving deworming treatment | 9 months
  The proportion of people in each village receiving deworming treatment was measured using household questionnaire surveys
proportion of dogs in each village receiving rabies vaccination | 9 months
  The proportion of dogs in each village receiving rabies vaccination was measured using household questionnaire surveys

SECONDARY OUTCOMES:
cost of delivery | 9 months
  the administration and delivery costs were measured
time people spent traveling | 9 months
  the time people spent traveling to the central point to receive deworming or vaccinations for their dogs was measured and compared between the integrated and non-integrated arms of the study
Comparison with the national school-based deworming program | 9 months
  The proportion of registered school children that received deworming treatment in the national school-based deworming program and the intervention delivered by the study was compared in ten primary schools

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Lankester F, Davis A, Kinung'hi S, Yoder J, Bunga C, Alkara S, Mzimbiri I, Cleaveland S, Palmer GH. An integrated health delivery platform, targeting soil-transmitted helminths (STH) and canine mediated human rabies, results in cost savings and increased breadth of treatment for STH in remote communities in Tanzania. BMC Public Health. 2019 Oct 28;19(1):1398. doi: 10.1186/s12889-019-7737-6. PMID 31660915